CLINICAL TRIAL: NCT00456339
Title: The Effect of a Combination of Systemic Steroids and Antibiotics on Obstructive Sleep Apnea Syndrome in Children
Brief Title: Systemic Steroids Plus Antibiotics in Sleep Apnea Syndrome in Children
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Problems recruiting; patient relapse following treatment
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 001 (14397A)
Record Dates: First submitted 2007-04-03; First posted 2007-04-04 (Estimated); Last update posted 2013-09-05 (Estimated); Status verified 2013-09

CONDITIONS: Obstructive Sleep Apnea Syndrome
Keywords: Obstructive sleep apnea syndrome (OSAS) in children
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Prednisolone; Amoxicillin; Clavulanic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Prednisolone and amoxicillin/clavulanate — Prednisolone 1mg/kg QD for 5 days Amoxicillin/clavulanate 45mg/Kg/d divided BID for 10 days

SUMMARY:
The purpose of this study is to investigate the effect of treatment with a steroid and antibiotic on the size of the tonsils and symptoms of children with OSAS.

DETAILED DESCRIPTION:
We will enroll children between 18 months and 12 years of age with mild sleep apnea and treat them with 5 days of prednisolone and 10 days of amoxicillin/clavulanate. We will obtain a questionnaire pre and post treatment and ask the parents to tell us if they think the child has improved enough after treatment to forego surgery. If not, they will undergo an adenotonsillectomy to relieve their sleep apnea and if yes, we will repeat the sleep study to make sure that the apnea has resolved.

ELIGIBILITY:
Inclusion Criteria:

* Polysomnogram results showing mild obstructive sleep apnea.

Exclusion Criteria:

* Significant medical problems
* Chronic medication intake (except bronchodilators and inhaled steroids)
* Allergy to penicillin or its derivatives.

Ages: 18 Months to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 4 (Actual)
Dates: Start 2006-07; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Sleep apnea questionnaire | 1-2 weeks post treatment
Size of tonsils | before and after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Fuad M Baroody, MD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States